CLINICAL TRIAL: NCT05048342
Title: A Multicenter, Open-label Phase 3 Study of Remibrutinib (LOU064) to Investigate the Safety, Tolerability and Efficacy for 52 Weeks in Adult Japanese Chronic Spontaneous Urticaria Patients Inadequately Controlled by H1-antihistamines
Brief Title: A Safety and Efficacy Study of Remibrutinib in the Treatment of CSU in Japanese Adults Inadequately Controlled by H1-antihistamines
Acronym: BISCUIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOU064A1301
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Bruton Tyrosine Kinase (BTK) inhibitor; Chronic Spontaneous Urticaria (CSU); Urticaria Activity Score (UAS); Weekly Urticaria Activity Score (UAS7); Hives Severity Score (HSS); Weekly Hives Severity Score (HSS7); Itch Severity Score (ISS); Weekly Itch Severity Score (ISS7); Angioedema Activity Score (AAS); Weekly Angioedema Activity Score (AAS7); Dermatology Life Quality Index (DLQI)
MeSH Terms: conditions — Chronic Urticaria | interventions — remibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LOU064 25 mg b.i.d. (Experimental): Patients were treated with remibrutinib 25 mg bis in die/twice a day (b.i.d.). LOU064 open-label treatment taken orally for 52 weeks.
  Interventions: Drug: LOU064

INTERVENTIONS:
Drug: LOU064 — Each patient took one film-coated tablet in the morning and one film-coated tablet in the evening (except the morning dose at the PK sampling visits, which were to be taken on site during the visit).
  Other Names: remibrutinib

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability and efficacy of remibrutinib (LOU064) in adult Japanese patients chronic spontaneous urticaria (CSU), who remain symptomatic despite treatment by H1-antihistamine (H1-AH) at locally label approved doses, for a duration of 52 weeks of treatment with remibrutinib and a post-treatment follow-up period of up to 4 weeks.

DETAILED DESCRIPTION:
The study consisted of three periods, the total study duration is up to 60 weeks: screening period of up to 4 weeks, open-label treatment period of 52 weeks (remibrutinib 25 mg b.i.d.), and a treatment free follow-up period of 4 weeks.

It was planned to include approximately 70 patients in the study; 71 patients were enrolled and included in the analyses.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent was required to be obtained prior to participation in the study.
* Male and female patients >= 18 years of age at the time of screening
* CSU duration for >= 6 months prior to screening (defined as the onset of CSU determined by the Investigator based on all available supporting documentation)
* Diagnosis of CSU inadequately controlled by second generation H1-AHs at the time of baseline (Day 1) defined as:

  * The presence of itch and hives for >= 6 consecutive weeks prior to screening despite the use of second generation H1-AHs during this time period
  * UAS7 score (range 0-42) >= 16, ISS7 score (range 0-21) >= 6 and HSS7 score (range 0-21) >= 6 during the 7 days prior to baseline (Day 1)
* Documentation of hives within three months before baseline (either at screening and/or at baseline; or documented in the patients' medical history)
* Willing and able to complete an UPDD for the duration of the study and adhere to the study protocol
* Patients were required to not have more than one missing UPDD entry (either morning or evening) in the 7 days prior to baseline (Day 1)

Exclusion criteria:

* Patients having a clearly defined predominant or sole trigger of their chronic urticaria (chronic inducible urticaria) including urticaria factitia (symptomatic dermographism), cold-, heat-, solar-, pressure-, delayed pressure-, aquagenic-, cholinergic-, or contact-urticaria
* Other diseases with symptoms of urticaria or angioedema, including but not limited to urticaria vasculitis, urticaria pigmentosa, erythema multiforme, mastocytosis, hereditary angioedema, or drug-induced urticaria
* Any other skin disease associated with chronic itching that might influence in the Investigator's opinion the study evaluations and results, e.g., atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus or psoriasis
* Evidence of clinically significant cardiovascular (such as but not limited to myocardial infarction, unstable ischemic heart disease, New York heart association Class III/IV left ventricular failure, arrhythmia and uncontrolled hypertension within 12 months prior to Visit 1), neurological, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic, hematological disorders, gastrointestinal disease or immunodeficiency that, in the Investigator's opinion, would compromise the safety of the patient, interfere with the interpretation of the study results or otherwise preclude participation or protocol adherence of the patient
* Significant bleeding risk or coagulation disorders
* History of gastrointestinal bleeding, e.g., in association with use of nonsteroidal anti-inflammatory drugs, that was clinically relevant (e.g., for which intervention was indicated or requiring hospitalization or blood transfusion)
* Requirement for anti-platelet medication, except for acetylsalicylic acid up to 100 mg/d or clopidogrel up to 75 mg/d. The use of dual anti-platelet therapy (e.g., acetylsalicylic acid + clopidogrel) is prohibited.
* Requirement for anticoagulant medication (for example, warfarin or Novel Oral Anti-Coagulants)
* History or current hepatic disease including but not limited to acute or chronic hepatitis, cirrhosis or hepatic failure or AST/ALT levels of more than 1.5 × ULN or International Normalized Ratio (INR) of more than 1.5 at screening

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Japan (12):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Urayasu, Chiba
  - Novartis Investigative Site, Izumiōtsu, Osaka
  - Novartis Investigative Site, Neyagawa, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Minato, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2425

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 13 centers in Japan.
Period: Overall Study
Arm/Group | LOU064 25 mg b.i.d.
Started (All enrolled patients were included in both the Full analysis set (FAS) and Safety set (SAF)) | 71
Completed | 68
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Subject decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | LOU064 25 mg b.i.d.
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (12.52)
Age, Customized [Number; unit: Participants]
  >= 18 and < 65 years | 66
  >= 65 and < 85 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 17
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
  Treatment emergent Adverse Event (TEAEs) in this study are events that started after the first dose of study treatment and until 30 days after the last study treatment, or events present prior to the first dose of treatment which increased in severity based on preferred term within 30 days after the last study treatment.
Time Frame: Baseline up to 30 days after last dose of study medication, assessed up to approximately 56 weeks
Population: Safety Set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25 mg b.i.d.
Number analyzed (Participants) | 71
Participants
  Subjects with at least one Adverse Event (AE) | 62
  Subjects with serious or other significant events - Death | 0
  Subjects with serious or other significant events - Non-fatal SAE(s) | 3
  Subjects with serious or other significant events - Discontinued study treatment due to any AE(s) | 1

2. Secondary Outcome: Mean Change From Baseline in Weekly Urticaria Activity Score (UAS7) at Week 12
Description: Change from Baseline in Weekly Urticaria Activity Score (UAS7) was assessed to evaluate the efficacy of Remibrutinib in Chronic Spontaneous Urticaria (CSU) patients. The Weekly Urticaria Activity Score (UAS7) is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the weekly UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | LOU064 25 mg b.i.d.
Number analyzed (Participants) | 71
Unit on a scale | -18.14 (10.992)

3. Secondary Outcome: Number of Participants Who Achieved Disease Activity Control (UAS7 =< 6) at Week 12
Description: The percentage of patients achieving disease activity control (UAS7 =< 6) at Week 12 was assessed to evaluate the efficacy of Remibrutinib in Chronic Spontaneous Urticaria (CSU) patients. The UAS7 is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25 mg b.i.d.
Number analyzed (Participants) | 71
Participants | 30

4. Secondary Outcome: Number of Participants Who Achieved Complete Absence of Hives and Itch (UAS7 = 0) at Week 12
Description: The proportion of patients achieving complete absence of hives and itch (UAS7 = 0) at Week 12 was assessed to evaluate the efficacy of Remibrutinib in Chronic Spontaneous Urticaria (CSU) patients. The UAS7 is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25 mg b.i.d.
Number analyzed (Participants) | 71
Participants | 15

5. Secondary Outcome: Change From Baseline in Weekly Itch Severity Score (ISS7) at Week 12
Description: The severity of the itch was recorded by the participant twice daily in their electronic Diary, on a scale of 0 (none) to 3 (severe). A weekly score (ISS7) was derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score was therefore 0 - 21 (highest itch severity).
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | LOU064 25 mg b.i.d.
Number analyzed (Participants) | 71
Unit on a scale | -8.01 (4.703)

6. Secondary Outcome: Change From Baseline in Weekly Hives Severity Score (HSS7) at Week 12
Description: The hives (wheals) severity score, defined by number of hives, was recorded by the participant twice daily in their electronic Diary, on a scale of 0 (none) to 3 (> 12 hives/12 hours). A weekly score (HSS7) was derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score was therefore 0 - 21 (highest hives activity).
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | LOU064 25 mg b.i.d.
Number analyzed (Participants) | 71
Unit on a scale | -10.12 (6.845)

7. Secondary Outcome: Number of Participants Who Achieved Early Onset of Disease Activity Control (UAS7 =< 6) at Week 2
Description: The percentage of patients achieving disease activity control (UAS7 =< 6) at Week 2 was assessed to evaluate the efficacy of Remibrutinib in Chronic Spontaneous Urticaria (CSU) patients. The UAS7 is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: Week 2
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25 mg b.i.d.
Number analyzed (Participants) | 71
Participants | 29

8. Secondary Outcome: Number of Participants Who Achieved Dermatology Life Quality Index (DLQI) = 0-1 at Week 12
Description: The Dermatology Life Quality Index (DLQI) is a 10-item (grouped in 6 domains) dermatology-specific quality of life (QoL) measure. Participants are rating their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives thinking about the previous 7 days. An overall score is calculated and ranges from 0 to 30 (higher score meaning worse disease-related QoL). Domain scores are calculated for: Symptoms and Feelings (0-6), Daily Activities (0-6), Leisure (0-6), Work and School (0-3), Personal Relationships (0-6), Treatment (0-3). The overall DLQI score range was split into score bands and validated in terms of their meaning/relevance to patients as follows: 0-1 (No effect on patient's life), 2-5 (Small effect on patient's life), 6-10 (Moderate effect on patient's life), 11-20 (Very large effect on patient's life), 21-30 (Extremely large effect on patient's life).
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25 mg b.i.d.
Number analyzed (Participants) | 71
Participants | 39

9. Secondary Outcome: Mean Cumulative Number of Weeks With Disease Activity Control (UAS7 =< 6) up to Week 12
Description: Maintaining disease activity control was assessed as cumulative number of weeks with an UAS7 =< 6 response between baseline and Week 12. The UAS7 is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: Up to Week 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | LOU064 25 mg b.i.d.
Number analyzed (Participants) | 71
Weeks | 4.6 (4.86)

10. Secondary Outcome: Mean Cumulative Number of Angioedema Occurrence-free Weeks (AAS7 = 0 Response) up to Week 12
Description: Angioedema occurrence was recorded once daily in the evening in the electronic Diary by the participant. Reporting the occurrence of angioedema was used as opening question for the assessment of the Angioedema Activity Score (AAS). The AAS consists of 5 questions with 4 answer options (scored 0-3) for each item, with a minimum score of 0 and a maximum score of 15 per day. The AAS score over 7 days (AAS7) ranges from 0 (no angioedema episodes) to 105 (highest angioedema severity).
Time Frame: Up to Week 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | LOU064 25 mg b.i.d.
Number analyzed (Participants) | 71
Weeks | 10.0 (3.63)

ADVERSE EVENTS:
Time Frame: On-treatment adverse events and deaths were reported from first dose of study medication up to 30 days after last dose of study medication, assessed up to approximately 56 weeks
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. The safety analysis were done on the safety population, which included all randomized subjects who received at least one dose of study medication.
Arm/Group | LOU064 25 mg b.i.d.
All-Cause Mortality (participants affected / at risk) | 0/71
Serious Adverse Events (participants affected / at risk) | 3/71
Other Adverse Events (participants affected / at risk) | 53/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LOU064 25 mg b.i.d. (N=71)
Meniere's disease (Ear and labyrinth disorders) | 1
Epiretinal membrane (Eye disorders) | 1
Rhegmatogenous retinal detachment (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LOU064 25 mg b.i.d. (N=71)
Diarrhoea (Gastrointestinal disorders) | 6
Pyrexia (General disorders) | 4
COVID-19 (Infections and infestations) | 14
Cystitis (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 7
Tonsillitis (Infections and infestations) | 5
Dyslipidaemia (Metabolism and nutrition disorders) | 4
Headache (Nervous system disorders) | 9
Acne (Skin and subcutaneous tissue disorders) | 5
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4
Eczema (Skin and subcutaneous tissue disorders) | 6
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 4
Purpura (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT05048342/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT05048342/SAP_001.pdf